CLINICAL TRIAL: NCT01377324
Title: In Vivo Imaging of the Effect of Fulvestrant on the Availability of Estrogen Receptor Binding Sites in Metastatic Breast Tumor Lesions Using FES-PET
Brief Title: Molecular Imaging of Fulvestrant Effects on Availability of ER Binding Sites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RUG2010-2611
Record Dates: First submitted 2011-05-19; First posted 2011-06-21 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Fulvestrant; FES; PET; Positron; Emission; Tomography; Fluoroestradiol; FES-PET; Molecular Imaging; Estrogen Receptor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Fluoroestradiol-PET is performed at baseline, after 1 month, and 3 months
  Interventions: Other: Diagnostic intervention: Positron Emission Tomography with 16-alpha-[18-fluoro]-17betaestradiol

INTERVENTIONS:
Other: Diagnostic intervention: Positron Emission Tomography with 16-alpha-[18-fluoro]-17betaestradiol — A FES-PET/(CT) will be performed thrice during protocol execution. Patients will be injected with ~200MBq 18F-FES

SUMMARY:
The dose of fulvestrant to optimally downregulate estrogen receptors (ER) is currently subject of debate. Effects of fulvestrant on the ERs may be evaluable by molecular imaging using positron emission tomography with the ER-specific FES tracer. In this pilot study we will evaluate the effects of the new dose of fulvestrant (500mg i.m.)on the availability of ER binding sites in 15 metastatic breast cancer patients.

DETAILED DESCRIPTION:
The estrogen receptor (ER) is expressed in approximately 70% of the breast carcinomas. In these patients signaling via the ER induces proliferation and cell survival of malignant cells. Fulvestrant can inhibit this signaling route by blocking the receptor and decreasing ER-expression by increasing its turn-over rate.

The historical standard dose of fulvestrant was 250mg every 28 days i.m.; however studies performing serial biopsies showed that ER-downregulation was suboptimal. Recently the standard dose has been set to 500mg i.m. on day 1; 14; 28 and every 28 days thereafter. Although slightly more effective than the 250mg dose, still questions remain with respect to the required dose to establish maximal downregulation of ER-signaling.

Immunohistochemistry only provides static information, i.e. the level of ER-expression. However, dynamic information evaluating the effects of fulvestrant on occupancy of ERs, may also be valuable.

Whole-body imaging of the availability of ER binding sites using FES-PET may prove valuable to evaluate the effects of fulvestrant on the ER non-invasively in individual patients. This potentially allows adjustment of dosing in individual patients to aid therapy efficacy.

In this pilot-study we will evaluate 15 metastatic breast cancer patients. All patients will undergo FES-PET/CT at baseline, FES-PET after 1 month, and FES-PET/CT after three months. Hormone- and fulvestrant levels will be measured in all patients. Whenever possible, tumor biopsies will be performed to correlate to FES-PET results.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with a history of histological proven ER-positive primary breast cancer and, whenever available, histological proven ER-positive recurrence. 2. Post-menopausal status (age ≥ 45 years with amenorrhea for > 12 months or prior bilateral ovariectomy 3. Documentation of a negative pregnancy test must be available for women less than 2 years after menopause 4. Progressive disease after 2 lines of hormonal therapy 5. No previous fulvestrant treatment 6. ER-antagonists should be discontinued for 5 weeks prior to FES-PET to prevent false negative FES-PET results. The use of aromatase inhibitors is allowed 7. ECOG performance status 0, 1 or 2 8. Life expectancy > 3 months 9. Creatinine clearance ≥ 30 ml/min 10. Age ≥ 18 years 11. Signed written informed consent 12. Able to comply with the protocol

Exclusion Criteria:

* 1. Evidence of central nervous system metastases 2. Presence of life-threatening visceral metastases 3. > 3 lines of endocrine therapy for metastatic disease 4. > 2 lines of chemotherapy in metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Visualize and quantify changes in FES uptake in tumor lesions during fulvestrant 500mg therapy | baseline; 1 month; 3 months
  FES-uptake will be calculated for all tumor lesions at baseline, 1 month and 3 months.
  Changes between FES-uptake during fulvestrant therapy will be calculated for:
  * 3 months minus baseline
  * 3 months minus 1 month
  * 1 month minus baseline
To evaluate the proportion of patients with an incomplete down-regulation/occupancy of ERs as determined by FES-PET | baseline, 1 month and 3 months
  FES-uptake will be calculated for all tumor lesions at baseline, after 1 month and after 3 months.
  Incomplete down-regulation/ occupancy of ERs is defined as 1) an absolute SUV> 1.5, and 2) a relative decrease in SUV of <75% during fulvestrant therapy.
  The proportion of patients that match these criteria will be given for:
  * 1 month minus baseline
  * 3 months minus baseline

SECONDARY OUTCOMES:
The feasibility to quantify changes in FES-uptake in liver metastases | baseline, 1 month and 3 months
  Liver metastases detected on PET/CT will be serially quantified at the 3 different time points to evaluate the feasibility to quantify liver lesions on FES-PET/CT
to correlate FES-PET results to patient and tumor response on fulvestrant therapy | baseline, 1 month, 3 months
  Patients will be categorized as responders and non-responders by standard follow-up (monthly visits, 3-monthly CT, other techniques when indicated).
  The predictive value of FES-PET for response to fulvestrant will be calculated for:
  * baseline FES-uptake
  * changes in FES-uptake from baseline to 1 month
  * changes in FES-uptake from baseline to 3 months
  Lesion-based evaluation will be performed for measurable lesions as defined by RECIST criteria, and changes in diameter will be correlated to changes in FES-uptake at:
  * 1 month minus baseline
  * 3 months minus baseline
Explorative analysis to correlate several factors (among which tumor burden, ER-expression, fulvestrant levels, estradiol levels, patient weight) to FES uptake will be performed. | baseline, 1 month and 3 months
  Explorative analysis to correlate several factors at different timepoints (baseline, 1 month, 3 months) to FES uptake.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Mortimer JE, Dehdashti F, Siegel BA, Trinkaus K, Katzenellenbogen JA, Welch MJ. Metabolic flare: indicator of hormone responsiveness in advanced breast cancer. J Clin Oncol. 2001 Jun 1;19(11):2797-803. doi: 10.1200/JCO.2001.19.11.2797. PMID 11387350
- [Background] Linden HM, Stekhova SA, Link JM, Gralow JR, Livingston RB, Ellis GK, Petra PH, Peterson LM, Schubert EK, Dunnwald LK, Krohn KA, Mankoff DA. Quantitative fluoroestradiol positron emission tomography imaging predicts response to endocrine treatment in breast cancer. J Clin Oncol. 2006 Jun 20;24(18):2793-9. doi: 10.1200/JCO.2005.04.3810. Epub 2006 May 8. PMID 16682724
- [Background] Howell A, Bergh J. Insights into the place of fulvestrant for the treatment of advanced endocrine responsive breast cancer. J Clin Oncol. 2010 Oct 20;28(30):4548-50. doi: 10.1200/JCO.2010.30.6266. Epub 2010 Sep 20. No abstract available. PMID 20855842